CLINICAL TRIAL: NCT05057403
Title: UK Imaging Diabetes Study Seeing Diabetes Clearly
Acronym: UKIDS
Status: Recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/WM/0007
Record Dates: First submitted 2021-09-01; First posted 2021-09-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, white blood cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes: Patients with type 2 diabetes, especially individuals who have been diagnosed in the last three years
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI is not part of Pathway for patient with type two diabetes.

SUMMARY:
Prospective, observational cohort study to cross-sectionally assess the health of multiple organs, using multiparametric abdominal magnetic resonance imaging (MRI) scan, and understand if resulting MRI metrics can predict future clinical events over a period of 5 years, in adult patients with type 2 diabetes lacking history of cardiovascular disease.

DETAILED DESCRIPTION:
This will be a multi-site study adopting a prospective, observational cohort study design. There will be no intervention to the standard of care. Study participants will be enrolled in this study for a total of 5 years, with only 1 month of active participation. Participants will be required to attend a screening visit and 2 study visits. The screening visit will involve a medical review and receiving informed consent based on the participant information leaflet already communicated to the patient, pre-screening. The first study visit- baseline (visit 1) - will involve anthropometric measurements and taking a blood and urine sample in order to perform standard of care measurements for type 2 diabetes at baseline and relevant circulating biomarkers. The second study visit will involve having a multi-organ, multiparametric MRI scan. Both visits will be within 28 days of the screening visit and carried out at local study sites.

MRI metrics of organ health, clinical outcome measurements, blood samples and urine samples will be collected to assess the natural history of diabetes disease progression. Participants will be asked to give consent for access to their medical records held at NHS England and, if available, at their local GP surgery or hospital. Medical records access will include Hospital admissions (Hospital Episode Statistics), and mortality data collected by the Office for National Statistics and provided by NHS England to meet the primary objective. This data will be collected at 1, 3 and 5 years after baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age and diagnosed with type 2 diabetes, with or without diabetic retinopathy.
* Participant willing and able to give informed consent for participation in the study.

Exclusion Criteria:

In 12 months prior to consent, evidence of existing cardiovascular event defined as at least one of:

* myocardial infarction
* ischaemic stroke
* hospital admission/discharge for unstable angina
* heart surgery
* unstable angina
* transient ischemic attack
* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (standard MR exclusion criteria including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Patients with known autoimmune hepatitis, viral hepatitis, Wilson's disease or known significant structural renal tract abnormality.
* Patients with known alcohol dependency.
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants, aged 18 years of age and over with type 2 diabetes lacking history of cardiovascular disease. Recruitment will be carried out from patients identified following diabetes or diabetic retinopathy diagnoses or via self-referral.
  1. Diabetes referral appointments
  2. Diabetic retinopathy referral appointments
  3. Primary care and diabetes clinics - including GP practices
  4. Participant Identification Centres
  5. Diabetes Eye Screening Programmes (DESP)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Baseline liver MR metrics on incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) in people with type 2 diabetes, without history of CV. | 3 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on cardiovascular clinical outcomes in a patient population with type 2 diabetes without history of cardiovascular disease.

SECONDARY OUTCOMES:
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death). | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death). | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death). | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of lower limb amputations | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of lower limb amputations | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of lower limb amputations | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of all-cause mortality | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of all-cause mortality | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of all-cause mortality | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of non-hepatic cancer | 1 year from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of non-hepatic cancer | 3 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
The effect of baseline liver MR metrics (cT1 and fat) on the incidence rate of non-hepatic cancer | 5 years from baseline
  The impact of liver fibroinflammation (cT1 from multi-organ MRI) on other diabetes-related outcomes
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase with incidence of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase with incidence of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite severe renal disease events (renal replacement therapy, renal death) | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite severe renal disease events (renal replacement therapy, renal death) | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite severe renal disease events (renal replacement therapy, renal death) | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite mild renal disease events (incident CKD, change in stage of CKD) | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite mild renal disease events (incident CKD, change in stage of CKD) | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of composite mild renal disease events (incident CKD, change in stage of CKD) | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of lower limb amputations | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of lower limb amputations | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of lower limb amputations | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of all-cause mortality | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of all-cause mortality | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of all-cause mortality | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of CV death, liver death, renal death, cancer death, other death | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of CV death, liver death, renal death, cancer death, other death | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of CV death, liver death, renal death, cancer death, other death | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension) | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of non-hepatic cancer | 1 year from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of non-hepatic cancer | 3 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
Potential effect of body composition, liver volume, and aortic (distensibility, diameter) MRI metrics increase and incidence of non-hepatic cancer | 5 years from baseline
  The impact that liver volume, whole body composition and, abnormalities in the aorta have on diabetes-related clinical outcomes using multiparametric MRI
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite severe renal disease events (renal replacement therapy, renal death) | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite severe renal disease events (renal replacement therapy, renal death) | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite severe renal disease events (renal replacement therapy, renal death) | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite mild renal disease events (incident CKD, change in stage of CKD) | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite mild renal disease events (incident CKD, change in stage of CKD) | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the composite mild renal disease events (incident CKD, change in stage of CKD) | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of the retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of lower limb amputations | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of lower limb amputations | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of lower limb amputations | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of all-cause mortality | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of all-cause mortality | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of all-cause mortality | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of non-hepatic cancer | 1 year from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of non-hepatic cancer | 3 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of retinopathy severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) on the incidence rate of non-hepatic cancer | 5 years from baseline
  The impact of the severity of diabetic retinopathy on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of 5-point MACE (CV death, non-fatal stroke, myocardial infarction, heart failure, hospitalisation for CV causes) | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death) | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death) | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite severe renal disease events (renal replacement therapy, renal death) | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of composite mild renal disease events (incident CKD, change in stage of CKD) | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of retinal intervention (photocoagulation, Vity, or use of anti-vascular endothelial growth factor injections) | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of lower limb amputations | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of lower limb amputations | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of lower limb amputations | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of all-cause mortality | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of all-cause mortality | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of all-cause mortality | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of CV death, liver death, renal death, cancer death, other death | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of liver events (decompensation, hepatocellular carcinoma diagnosis, transplant, portal hypertension | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of non-hepatic cancer | 1 year from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of non-hepatic cancer | 3 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
The effect of age of T2DM diagnosis (early onset and under 45 year of age, usual onset) on the incidence rate of non-hepatic cancer | 5 years from baseline
  The impact of age of onset of T2DM on cardiovascular and other diabetes-related outcomes
Prevalence of patients with evidence of metabolic dysfunction-associated steatotic liver disease in patients with diabetic retinopathy of different severity (no DR, mild NPDR, moderate NPDR, severe NPDR, PDR, advanced PDR) | 1 year from baseline
  The co-prevalence of diabetic retinopathy (DR) and metabolic dysfunction-associated steatotic liver disease (MASLD), using multi-parametric abdominal MRI
Correlations between liver MRI metrics (organ volume, fat infiltration and fibroinflammation) and eye metrics (retinal layer thickness by OCT, discrete retinopathy scores) | 1 year from baseline
  The correlation between severity of eye disease and MRI-derived metrics of liver disease using multiparametric MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Pattanshetty, Principal Investigator — Perspectum
Locations (12):
- United Kingdom (12):
  - Woodlands Medical Centre, Didcot, Oxfordshire
  - Eynsham Medical Centre, Eynsham, Oxfordshire
  - White Horse Medical Practice, Farringdon, Oxfordshire
  - Windrush Medical Practice, Witney, Oxfordshire
  - The House Partnership, Redhill, Surrey
  - Swansea Bay University Health Board, Baglan, Swansea
  - University Hospitals of Liverpool Group, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - The Manor Group, Oxford
  - Hedena Health, Oxford
  - St Bartholomew and Hollow Way Medical Practice, Oxford
  - Oxford Community Diagnostic centre, Oxford

IPD SHARING:
Plan to Share IPD: No